CLINICAL TRIAL: NCT01745523
Title: "Impact of Using Hydroxypropyl Cellulose (HPC) and Trehalose for Oocyte Vitrification in an Ovum Donation Program"
Brief Title: Use of a Synthetic Macromolecule (Hydroxypropyl Cellulose ) and Trehalose as Additives for Oocyte Vitrification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Ana Cobo, Cryobiology Unit Director at IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1206-C-103-AC; ClinicalTrials.gov (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2012-11-29; First posted 2012-12-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: Oocyte vitrification; survival rate; egg banking; ovum donation
MeSH Terms: conditions — Infertility | interventions — Trehalose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrified oocytes using HPC+Trehalose (Experimental): Oocytes are vitrified using the synthetic macromolecule HPC and trehalose
  Interventions: Procedure: Synthetic macromolecule HPC and trehalose
- Vitrified oocytes using SSS+ Sucrose (Active Comparator): Oocytes are vitrified using the SSS containing HSA and sucrose
  Interventions: Procedure: SSS containing HSA and sucrose

INTERVENTIONS:
Procedure: Synthetic macromolecule HPC and trehalose — Oocytes are vitrified using the synthetic macromolecule HPC and trehalose
  Arms: Vitrified oocytes using HPC+Trehalose
Procedure: SSS containing HSA and sucrose — • Oocytes are vitrified using the SSS containing HSA and sucrose
  Arms: Vitrified oocytes using SSS+ Sucrose

SUMMARY:
This study is aimed to evaluate the use of Hydroxypropyl Cellulose (HPC) as substitute for the traditional protein supplement (Synthetic Serum Substitute; SSS) and Trehalose as substitute for the most widely used sugar (Sucrose) in the vitrification solutions employed for oocyte vitrification.

DETAILED DESCRIPTION:
Vitrification involves the transformation of an aqueous solution into a very viscous solid avoiding ice formation. To achieve this, the vitrification protocols include high concentrations of cryoprotectants dissolved in a base medium supplemented with serum rich in protein. Traditionally available preparations contains human albumin (HSA). The most commonly used in vitrification solutions is the synthetic serum replacement (SSS) consisting of synthetic glycoporoteins and HSA. The replacement of human albumin by other fully synthetic components enables compliance with the European directives for classification of Class III medical device in accordance with the Manual for the Classification of Medical Devices in the regulatory framework of the European community, and therefore these media have the European CE conformity marking (Directive 93/42/EEC). According to European regulations, Class III medical devices are subject to special supervision and require certification exam or design type examination by a notified body. Commercial media supplied by Kitazato supplies ® (Tokyo, Japan) to be used in this study have been submitted to the whole process of evaluation and certification by the notified body BSI0086. Because of physical properties of hydroxypropyl cellulose (HPC), fully synthetic macromolecule, including the ability to form a viscous gel at low temperatures, this macromolecule has been proposed as a substitute for human origin albumin (HSA). Another necessary component of vitrification media is sucrose, which acts as an osmotic agent. Trehalose, a disaccharide present in nature is used by certain species to survive extreme conditions, being able to remain vitrified for years. This sugar has also been employed previously in cryobiology in some vitrification protocols. We have tested HPC and threhalose for oocytes vitrification in a pilot study, showing that no impairment in the survival rates, embryo development and pregnancy rates. The current study is a prospective randomized trial aimed to assess the outcome of ovum donation cycles conducted with vitrified oocytes using HPC and trehalose versus oocytes vitrified using traditional available solutions containing HAS and sucrose.

ELIGIBILITY:
Inclusion Criteria:

Donors:

* < 35 years old
* Normal physical and gynecological examinations
* No family history of hereditary or chromosomal diseases.
* Normal karyotype
* Negative screening for sexually transmitted diseases.

Oocyte recipients:

* Oocyte recipients < 50 years old
* Body mass index< 30
* < 2 previous IVF failures
* No severe male factor
* No recurrent miscarriage
* No hidrosalpinx
* No myoma
* No adenomyosis
* No AMH alterations

Exclusion Criteria:

Donors and recipients not meeting inclusion criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Survival after oocyte vitrification using cryoprotective solutions containing hiroxipropilcelulosa (HPC) and trehalose. | >2 hours
  After warming and embryo transfer. Survival will be evaluated morphologically two hours after warming.

SECONDARY OUTCOMES:
Embryo development | From time of thawing until pregnancy outcome (0-9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cobo, PhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain